CLINICAL TRIAL: NCT05489055
Title: Department of Radiology
Brief Title: Effects of Contrast Media Temperature on Image Quality and Clinical Adverse Events in Coronary CTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Emergency Medical Center (Other)
Collaborators: Army Medical Center of PLA (Other Government)
Responsible Party: Principal Investigator, Hao Wu, Associate professor, Chongqing Emergency Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChongqingEMC
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Contrast Media Adverse Reaction
Keywords: Computed Tomography Angiography; Low-osmolality contrast media; Image quality; Clinical adverse event
MeSH Terms: interventions — Iopamidol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBT-CM (basic body temperature) group (Experimental): BBT-CM (basic body temperature) group received contrast media warmed to body temperature (37°C[99°F]) before coronary CTA.
  Interventions: Drug: Iopamidol
- RT-CM (room temperature) group (Active Comparator): RT-CM (room temperature) group received contrast media at room temperature (~23°C [~73°F]) before coronary CTA.
  Interventions: Drug: Iopamidol

INTERVENTIONS:
Drug: Iopamidol — A contrast bolus of iopamidol-370 (370 mg I/ml) (iopamidol injection; Consun Pharmaceutical, China) was injected at a ﬂow rate of 4.5-6 mL/s through an 18-20-gauge intravenous antecubital catheter by using a power injector (Ulrich, Germany). The total dose of iopamidol-370 was approximately 0.9 ml /kg body weight.

SUMMARY:
Extrinsic prewarming of iodinated CT contrast media (CM) to body temperature reduces viscosity and injection pressures. However, guideline recommendations on the necessity to prewarm iodinated CM are conflicting. And studies examining the effect of extrinsic warming CM for coronary CTA(CCTA) on clinical adverse events and image quality are lack.

Enrolled patients of chest pain or coronary artery disease screening were eligible for this a double-blinded, randomized noninferiority trial, and equally allocated into two group randomly: BBT-CM (basic body temperature) group received 37°C CM; RT-CM (room temperature) group received ~23°C CM. A state-of-the-art individualized CM (iopamidol at 370 mg I/mL) injection protocol was used, based on body weight.

ELIGIBILITY:
Inclusion Criteria:

* Coronary symptomatic patients (i.e., chest pain).
* Patients for Coronary artery disease screening

Exclusion Criteria:

* Hemodynamic instability
* Renal insufficiency (estimated glomerular filtration rate <30 mL/min per 1.73 m2)
* Prior adverse reactions to iodinated CM
* Age younger than 18 years
* Inability to place an 18-gauge needle.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Vessel Attenuation | Expected within one month after the coronary CTA is performed
  Mean attenuation in Hounsfield Units (HU) is based on coronary bifurcation, preferably right coronary artery (RCA), left anterior descending artery (LAD), and left circumflex coronary artery (LCX)). Absolute difference in mean attenuation of coronary vessels between groups was calculated with a two-sided 95% confidence interval of the difference.

SECONDARY OUTCOMES:
Allergic or allergiclike reaction | 30 minutes after coronary CTA
  Allergic and allergic-like reactions were identified by evaluating notes within the EMR for elements of such reactions specified in nomenclature from the ACR manual. Allergic reactions were recorded according to symptoms of an immune response to the CM, such as feeling cold urticaria or pruritis.
Extravasations | Expected during the coronary CTA scan.
  The radiology staff recorded an estimate of the volume of extravasated contrast media
Objective image quality - Signal-to-noise ratio(SNR) | Within one month after the CT is performed
  mean attenuation of vessel divided by the mean SD
Objective image quality -Contrast-to-noise ratio(CNR) | Within one month after the CT is performed
  mean vascular attenuation minus HU of the vessel, divided by the SD of the attenuation of epicardial fat surrounding left main coronary artery and then divided by image noise
CT Dose Index (CTDI)vol | Expected during the coronary CTA is performed
  CTDIvol (in mGy) the patient received
Physiologic reactions-Urgency desire | Immediately after CT
  Urgency desire is defined in the questionnaire as the sudden and intense ''urge'' or need to urinate and scored 1=Not at all, 2=A little, 3= Moderately, 4=A great deal, and 5=A very great deal.
Body Mass Index | Right before the scan is performed
  The formula is BMI = kg/m2 , where kg is a person's weight in kilograms and m2 is their height in metres squared.
Subjective image quality | Within one month after the CT is performed
  Rated in consensus on a 5-point Likert scale by two radiologists: 1=excellent (absence of artifacts related to motion or coronary calcification); 2=good (minor artifacts); 3=moderate (considerable artifacts but maintained visualization of the arterial lumen); and 4=poor (non-diagnostic because of severe motion artifacts or severe coronary calcification).
Heart rate | During the coronary CTA.
  Heart rate (beats per minute) is monitor during the coronary CTA.
Flow rate | Within one month after the CT is performed
  Flow rate of the contrast media in ml/s.
Dose-length product (DLP) | Within one month after the CT is performed
  DLP (in mGycm) the patient received

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Emergency Mediacl Centre, Chongqing, Chonqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basharat NF, Ranganathan K, Kang PT, Gridley DG, Roh AT. Effect of Extrinsic Warming of Low-Osmolality CT Contrast Media (Iohexol 350) on Extravasations and Patient Reaction Rates: A Retrospective Study. AJR Am J Roentgenol. 2022 Jan;218(1):174-179. doi: 10.2214/AJR.21.26256. Epub 2021 Jul 28. PMID 34319163
- [Result] Martens B, Wildberger JE, Van Kuijk SMJ, De Vos-Geelen J, Jeukens CRLPN, Mihl C. Influence of Contrast Material Temperature on Patient Comfort and Image Quality in Computed Tomography of the Abdomen: A Randomized Controlled Trial. Invest Radiol. 2022 Feb 1;57(2):85-89. doi: 10.1097/RLI.0000000000000807. PMID 34280944
- [Derived] Peng C, Liu Y, Zhang H, Xu G, He C, Jian D, Liu H, Li C, Zeng P, Wu H. Effects of extrinsically warmed contrast media on image quality and clinical adverse events in patients undergoing coronary computed tomography angiography: a randomized controlled trial. Quant Imaging Med Surg. 2026 Jan 1;16(1):13. doi: 10.21037/qims-2025-121. Epub 2025 Dec 31. PMID 41521999